CLINICAL TRIAL: NCT03857646
Title: The Effect of Lipid Emulsions on Free Fatty Acids and Free Bilirubin in Premature Newborns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Meredith Collins, Physician, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-18-1000
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Prematurity
Keywords: parenteral nutrition; lipid emulsion; free bilirubin; free fatty acids
MeSH Terms: conditions — Premature Birth; Hyperphagia | interventions — soybean oil, phospholipid emulsion; Lipids

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intralipid (Other)
  Interventions: Drug: Intralipid, 20% Intravenous Emulsion
- Soybean oil Medium-chain triglycerides Olive oil Fish Oil (SMOF) lipid (Other)
  Interventions: Drug: Soybean oil Medium-chain triglycerides Olive oil Fish Oil (SMOF) lipid

INTERVENTIONS:
Drug: Intralipid, 20% Intravenous Emulsion — Lipids start at 1 g/kg/day and advance by 1 g/kg/day to a maximum of 3 g/kg/day as tolerated by the the neonate.
  Arms: Intralipid
Drug: Soybean oil Medium-chain triglycerides Olive oil Fish Oil (SMOF) lipid — Lipids start at 1 g/kg/day and advance by 1 g/kg/day to a maximum of 3 g/kg/day as tolerated by the the neonate.
  Arms: Soybean oil Medium-chain triglycerides Olive oil Fish Oil (SMOF) lipid

SUMMARY:
The goal of this research study is to compare the levels of free fatty acids and free bilirubin between two intravenous lipid emulsion products in premature newborns.

ELIGIBILITY:
Inclusion Criteria:

* premature newborns (<32 weeks gestation, stratified <28 weeks versus >28 weeks) <8 days of age
* receiving lipid infusions <1 g/kg/day at enrollment
* anticipated to be treated with 3 g/kg/day for a minimum of 48 hours.

Exclusion Criteria:

* patients with direct hyperbilirubinemia >1.5 mg/dl
* with suspected sepsis meeting Systemic inflammatory response syndrome (SIRS) criteria
* undergoing treatment with a continuous infusion of morphine
* with a continuous infusion of pressors (dopamine, dobutamine, epinephrine, etc.)
* positive blood cultures

Ages: 0 Days to 8 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-03-02 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cody Arnold, MD, Study Director — UT Houston HSC
Locations (1):
- University Texas Houston HSC, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intralipid | Soybean Oil Medium-chain Triglycerides Olive Oil Fish Oil (SMOF) Lipid
Started | 33 | 33
Completed One Day of Infusion at 3 g/kg/Day | 31 | 29
Completed Two Days of Infusion at 3 g/kg/Day | 29 | 25
Completed | 29 | 25
Not Completed | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- SMOF Lipid: SMOF lipid: Lipids start at 1 g/kg/day and advance by 1 g/kg/day to a maximum of 3 g/kg/day as tolerated by the the neonate.
- Total: Total of all reporting groups
Arm/Group | Intralipid | SMOF Lipid | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: days] — Population: Data was not collected for one participant in the Intralipid arm. Data was not collected for one participant in the SMOF lipid arm.
  days
    number analyzed (Participants) | 32 | 32 | 64
    (all) | 1.81 (0.53) | 1.83 (0.37) | 1.82 (0.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 15 | 15 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Free Bilirubin (UB) Serum Levels
Time Frame: first day of infusion at 3 g/kg/day
Population: UB levels were measured in 2/3 of the samples before the pandemic closed the analytic laboratory, and the other 1/3 were assessed post-pandemic 1.5 years later. The UB data are invalid due to an issue associated with the delay, that is, the UB measurement device developed by the bench scientist colleagues was recalibrated in the interim such that the UB results pre vs post recalibration are incomparable.
  Data were not collected for 1 participant in the Intralipid arm.
Measure: Mean (Standard Deviation); unit: Nanomoles/Liter (nM)
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 30 | 29
Nanomoles/Liter (nM) | 10.5 (7.5) | 9.4 (7.0)

2. Primary Outcome: Free Bilirubin (UB) Serum Levels
Time Frame: second day of infusion at 3 g/kg/day
Population: UB levels were measured in 2/3 of the samples before the pandemic closed the analytic laboratory, and the other 1/3 were assessed post-pandemic 1.5 years later. The UB data are invalid due to an issue associated with the delay, that is, the UB measurement device developed by the bench scientist colleagues was recalibrated in the interim such that the UB results pre vs post recalibration are incomparable.
Measure: Mean (Standard Deviation); unit: Nanomoles/Liter (nM)
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 29 | 25
Nanomoles/Liter (nM) | 10.2 (7.8) | 7.4 (2.2)

3. Secondary Outcome: Unbound Free Fatty Acid (FFAu) Serum Level
Description: To measure unbound free fatty acid level, a fluorescent probe called Acrylodan-Labeled Intestinal Fatty Acid Binding Protein 2 (ADIFAB2) was used. The ADIFAB2 fluorescent probe is a fatty acid binding protein complexed with a fluorescent group. Once mixed with a sample, the ADIFAB2 fluorescent probe binds all unbound free fatty acid in the sample; therefore, measurement of fluorescence indicates the amount of unbound free fatty acid in the sample. After binding of the ADIFAB2 fluorescent probe to the sample, fluorescence intensities are measured at two wavelengths (550 nanometers and 457 nanometers), and for this outcome measure the R value is reported. The R value is the ratio of the fluorescence intensity at 550 nanometers to the fluorescence intensity at 457 nanometers.
Time Frame: first day of infusion at 3 g/kg/day
Population: FFAu levels were measured in 2/3 of the samples before the pandemic closed the analytic laboratory, and the other 1/3 were assessed post-pandemic 1.5 years later. The FFAu data are invalid due to an issue associated with the delay, that is, there was severe sample degradation of the FFAu samples that were measured post-pandemic due to prolonged freezing and refreezing-rethawing.
Measure: Mean (Standard Deviation); unit: ratio value (R)
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 31 | 29
ratio value (R) | 0.112 (0.034) | 0.106 (0.008)

4. Secondary Outcome: Unbound Free Fatty Acid (FFAu) Serum Level
Description: To measure unbound free fatty acid level, a fluorescent probe called ADIFAB2 was used. The ADIFAB2 fluorescent probe is a fatty acid binding protein complexed with a fluorescent group. Once mixed with a sample, the ADIFAB2 fluorescent probe binds all unbound free fatty acid in the sample; therefore, measurement of fluorescence indicates the amount of unbound free fatty acid in the sample. After binding of the ADIFAB2 fluorescent probe to the sample, fluorescence intensities are measured at two wavelengths (550 nanometers and 457 nanometers), and for this outcome measure the R value is reported. The R value is the ratio of the fluorescence intensity at 550 nanometers to the fluorescence intensity at 457 nanometers.
Time Frame: second day of infusion at 3 g/kg/day
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio value (R)
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 29 | 25
ratio value (R) | 0.105 (0.008) | 0.105 (0.008)

5. Secondary Outcome: Free Fatty Acid (Total) Serum Level
Time Frame: second day of infusion at 3 g/kg/day
Population: Data were not collected for this outcome measure.
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Direct Bilirubin >1.8 Milligrams Per Deciliter (mg/dL)
Time Frame: first and/or second days of infusion at 3 g/kg/day
Population: Data are reported for all who had 1 or 2 days of infusion of 3 g/kg/day.
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 31 | 29
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Peak Serum Triglyceride Level >350 mg/dl
Time Frame: first or second days of infusion at 3 g/kg/day
Population: Of those who had 1 or 2 days of infusion of 3 g/kg/day, data were not collected for 1 participant in the Intralipid arm, and data were not collected for 2 participants in the SMOF lipid arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 30 | 27
Participants | 1 | 2

8. Secondary Outcome: Mean Serum Triglyceride Level
Time Frame: first day of infusion at 3 g/kg/day
Population: Of those who had infusion of 3 g/kg/day on the first day, data were not collected for 1 participant in the Intralipid arm, and data were not collected for 2 participants in the SMOF lipid arm.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 30 | 27
milligrams per deciliter (mg/dL) | 177.23 (91.73) | 139.37 (74.63)

9. Secondary Outcome: Mean Serum Triglyceride Level
Time Frame: second day of infusion at 3 g/kg/day
Population: Of those who had infusion of 3 g/kg/day for two days, data were not collected for 14 participants in the Intralipid arm, and data were not collected for 13 participants in the SMOF arm.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Intralipid | SMOF Lipid
Number analyzed (Participants) | 15 | 12
milligrams per deciliter (mg/dL) | 153.53 (63.84) | 159.5 (120.23)

ADVERSE EVENTS:
Time Frame: about 5 days
Arm/Group | Intralipid | SMOF Lipid
All-Cause Mortality (participants affected / at risk) | 2/33 | 1/33
Serious Adverse Events (participants affected / at risk) | 2/33 | 1/33
Other Adverse Events (participants affected / at risk) | 0/33 | 1/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralipid (N=33) | SMOF Lipid (N=33)
Death (General disorders) | 2 (2) | 1 (1)
Severe intraventricular hemorrhage (IVH) (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intralipid (N=33) | SMOF Lipid (N=33)
Received vasopressors to treat low blood pressure (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
UB and FFAu levels were measured in 2/3 of the samples before the pandemic, and the other 1/3 were assessed post-pandemic 1.5 years later. The UB and FFAu data are invalid due to 2 issues associated with the delay: (1) the UB measurement device was recalibrated in the interim such that the UB results pre vs post recalibration are incomparable and (2) for FFAu, there was severe sample degradation of the samples measured post-pandemic due to prolonged freezing and refreezing-rethawing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT03857646/Prot_SAP_000.pdf